CLINICAL TRIAL: NCT03973606
Title: Assessment of the Health Literacy Among Arab Women in East Jerusalem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HMO007819
Record Dates: First submitted 2019-05-23; First posted 2019-06-04 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Health Literacy; Cardiovascular Diseases
Keywords: Health literacy; East Jerusalem; Focus groups; Arabic Women
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: A 4-sessions workshop to improve health literacy among Arab women in Israel, with pre-post evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arab Women health literacy focus groups (No Intervention): Arab women in East Jerusalem will be part of focus groups. During the focus groups, a set of pre-prepared questions will be presented to the participants. The focus groups will be recorded and analyzed verbatim.
- Health literacy workshop (Experimental): Women from East-Jerusalem and other Arab communities in Israel will be invited to participate in a 4-sessions workshop designed to improve health literacy, self-efficacy when interacting with their physician and increase their cardiovascular health knowledge.
  Interventions: Other: Heath literacy assessment in Arab women in East Jerusalem

INTERVENTIONS:
Other: Heath literacy assessment in Arab women in East Jerusalem — A 4-sessions intervention to increase the participant's self-efficacy when interacting with their physician and increase their cardiovascular health knowledge.
  Other Names: Health literacy workshop
  Arms: Health literacy workshop

SUMMARY:
This is a two-stage study: The objective of the first stage is to explore health literacy (HL) needs and preferences of Arab women through conducting Focus Group Discussions (FGDs).

The second stage will employ conducting a HL intervention tailored to the participants' needs and preferences as presented in the FGDs. Objectives include increasing the percentage of women who utilize patient-doctor communication skills and increasing their cardiovascular disease (CVD) knowledge.The intervention consists of four sessions that will be conducted in municipality-sponsored women's groups in Jerusalem and other Arab communities. Questionnaires will be completed before and three months after the intervention. The study answers the following: Can HL workshops improve patient-doctor communication skills and CVD knowledge in Arab women.

DETAILED DESCRIPTION:
Arab women in Israel are at high risk of low health literacy due to lower levels of education and low socio-economic status. Health literacy (HL) refers to the skills and competencies enabling people to obtain and interpret health information and apply their knowledge to inform health-related decision-making. It's also defined as "the degree to which individuals have the capacity to obtain, understand, and process basic health information and services needed to make appropriate health decisions".

The objective of the first stage of the study is to explore health literacy needs and preferences of Arab women through conducting Focus Group Discussions (FGDs) with women in East Jerusalem. Six different focus groups will be conducted at three of the six municipality community centers in East Jerusalem. Participants will be recruited through identified community centers.

Each group will meet once for up to two hours. The study will be explained to them by an investigator who has been trained in the administration of focus groups, and they will be asked to sign a consent form. Discussions will be recorded without the names of the participants (they will be instructed not to use their names once the recording begins). At the end of the meeting, each participant will receive a bag and pamphlets with information regarding women's health.

The second stage will employ conducting a HL intervention tailored to the participants' needs and preferences as presented in the FGDs. Objectives include increasing the percentage of women who utilize patient-doctor communication skills and increasing their cardiovascular disease (CVD) knowledge.The intervention consists of four sessions that will be conducted in municipality-sponsored women's groups in Jerusalem and other Arab communities. Questionnaires will be completed before and three months after the intervention. The study answers the following: Can HL workshops improve patient-doctor communication skills and CVD knowledge in Arab women.

ELIGIBILITY:
Inclusion Criteria:

* All women aged 18-85 that attend and participate in the community's women's groups
* They must speak Arabic

Exclusion Criteria:

* Not in the age range of 18-85.
* Do not speak Arabic.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
assessment of health literacy level and elucidate factors that will improve health literacy (barriers, incentives, etc.…) among Arab women in East Jerusalem | within 6 months
  The assessment will be done through conduction of focus groups. Focus groups will be audio- recorded, transcribed and analyzed using Systematic text condensation, a descriptive and explorative analysis strategy. Which consists of four steps: 1) total impression - from chaos to themes; 2) identifying and sorting meanings units - from themes to codes; 3) condensation - from code to meaning; 4) synthesizing - from condensation to descriptions and concepts. It is expected that six focus groups will be sufficient to achieve saturation of themes. If results are not sufficient, investigators will ask to increase the number of focus groups.
Change in cardiovascular disease knowledge | At baseline and three months after intervention
  A self report questionnaire based on the American Heart Association's Cardiovascular, and assess the knowledge regarding heart attack symptoms, by answering yes/no to each item.
Change in perceived efficacy in patient-physician interaction | At baseline and three months after intervention
  Will be assessed using the 10-item Perceived Efficacy in Patient-Physician Interaction (PEPPI) (Maly, Frank, Marshall, Diametteo, Reuben, 1998). Participants respond to each question on a scale of 1 to 10, with 10 representing "very confident,'' and 1 representing "not at all confident". Higher scores represent positive outcome.
Change in remembering doctor's recommendations and reading blood test results | At baseline and three months after intervention
  A 2-item version derived from the Perceived Efficacy in Patient-Physician Interaction (PEPPI). Participants respond to each question on a scale of 1 to 5, with 5 representing "very confident,'' and 1 representing "not at all confident". Higher scores represent positive outcome.
change in health literacy | At baseline and three months after intervention
  Will be assessed using the Health Literacy Survey-Europe-Q16 (HLS-EU-Q16) a 16 question research instrument adapted for use in Israel. Participants respond to each question on a scale of 1 to 4, with 4 representing "fairly easy,'' and 1 representing "very difficult". Higher scores represent positive outcome.
Change in preparation for doctor's visit | At baseline and three months after intervention
  A 6-item questionnaire represents preferred actions that participant\pants do before their doctor appointment. The more items are selected, the higher the score is, hence representing a positive outcome.

SECONDARY OUTCOMES:
Change in Self-Rated Status of Health (SRH) | At baseline and three months after intervention
  A validated single item health measure in which participants rate the current status of their own health on a five-point scale, from excellent to poor
Change in perceived efficacy in reading and understanding the instruction for taking medications | At baseline and three months after intervention
  Participants will be asked "how confident do you feel you are able to follow the instructions on the label of a medication bottle?"

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD MPH, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Beit-Safafa community center, Jerusalem, Israel

REFERENCES:
- [Background] Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. J Am Geriatr Soc. 1998 Jul;46(7):889-94. doi: 10.1111/j.1532-5415.1998.tb02725.x. PMID 9670878